CLINICAL TRIAL: NCT01702779
Title: Nasal Humidified High Flow Oxygen During Weaning From Mechanical Ventilation : Ultrasonography Study
Acronym: HiFloLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Pitié-Salpêtrière Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0107
Record Dates: First submitted 2012-04-24; First posted 2012-10-08 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Adult Patients Ventilated More Than 48 h; Stable Respiratory and Hemodynamic Conditions for SBT; Consent of Patients; Arterial Line
Keywords: Weaning from mechanical ventilation; Lung ultrasound; Oxygen inhalation therapy
MeSH Terms: interventions — Respiration, Artificial

ARMS (2):
- optiflow (Other)
  Interventions: Other: mechanical ventilation
- O2 (Other)
  Interventions: Other: mechanical ventilation

INTERVENTIONS:
Other: mechanical ventilation — Prospective, randomized clinical multicentric study in ICU (Intensive Care University)during weaning from mechanical ventilation.
  Arms: optiflow
Other: mechanical ventilation — Prospective, randomized clinical multicentric study in ICU (Intensive Care University)during weaning from mechanical ventilation.
  Arms: O2

SUMMARY:
This is a prospective, randomized clinical multicentric study in ICU (Intensive Care University)during weaning from mechanical ventilation.

DETAILED DESCRIPTION:
Prospective randomized clinical multicentric study on ICU (Intensive Care University) comparing nasal humidified high flow therapy versus standard oxygen with Lung Ultrasound Score during weaning from mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ventilated more than 48 h
* Stable respiratory and hemodynamic conditions for SBT
* Consent of patients
* Arterial line

Exclusion Criteria:

* COBP
* Laryngeal dyspnea
* Tracheostomy
* Arythmya
* No echogenicity
* Paraplegia >T8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
variations of lung ultrasound score | 24 hours after extubation

SECONDARY OUTCOMES:
Lung ultrasound score | at baseline, 4-6 hours after extubation, 24 hours after extubation, 48 hours after extubation
rates of patients with postextubation distress | during the 48th post-extubation
Electrical Impedance tomography | at baseline, 4-6 hours after extubation, 24 hours after extubation, 48 hours after extubation
Epithelial and endothelial biomarkers | at baseline, 4-6 hours after extubation, 24 hours after extubation, 48 hours after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France